CLINICAL TRIAL: NCT03937674
Title: Heart Steps: Adaptive mHealth Intervention for Physical-Activity Maintenance
Brief Title: An mHealth Mobile Application Supporting Maintenance of Physical Activity Among Men and Women With High Blood Pressure
Acronym: HeartSteps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of Michigan (Other); University of California, San Diego (Other); Harvard University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1257484
Record Dates: First submitted 2019-04-24; First posted 2019-05-06 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Physical Activity
Keywords: Physical Activity; Mobile Health; Self Monitoring; Wearable Sensors; Tailored Health Communication; Implementation Intentions; Mobile Apps; Anti-Sedentary Behavior; Opportunistic Physical Activity; Health Belief Model
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: At each "decision time"-a time point when an intervention component can be delivered-each day of the study each participant is randomized between intervention or no intervention (delivery of a contextually tailored activity suggestion or no suggestion; morning motivational message or no motivational message)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HeartSteps Intervention (Experimental): For activity suggestions, at each available decision time, each participant is randomly assigned to either receive an activity suggestion or not.
  Interventions: Behavioral: HeartSteps: A just-in-time intervention for increasing physical activity among sedentary adults.

INTERVENTIONS:
Behavioral: HeartSteps: A just-in-time intervention for increasing physical activity among sedentary adults. — HeartSteps is a smartphone based mHealth intervention that contains the following intervention components: (1) contextually-tailored suggestions for activity; (2) motivational messages aimed at keeping individuals motivated to be active; (3) planning of the next week's activity; and (4) adaptive weekly activity goals. Activity suggestions provide individuals with suggestions for how they can be active, and are tailored based on time of day, user's location, day of the week (weekend/weekday), and weather. Motivational messages are delivered to individuals via a push notification. Activity planning asks users to create a plan of how they will be active in the coming week. Participants are prompted to plan once a week. Each week, as part of the weekly planning, HeartSteps suggests an activity goal for the coming week based on their activity levels the previous week. Participants can edit the suggested goal, and the system-suggested goals top out at 150 minutes of activity per week.

SUMMARY:
The aim of this research is to evaluate the efficacy of contextually tailored activity suggestions and activity planning for increasing physical activity among sedentary adults.

DETAILED DESCRIPTION:
This project file refers to Aim 2 and Aim 3 of the National Heart, Lung, and Blood Institute (NHLBI) grant. Aim 1 is registered in clinical trials.gov under a separate project file number, NCT03225521.

Many of the risk factors for heart disease are behavioral, such as physical inactivity, smoking, and diets high in saturated and trans-fats. Prevention programs are effective at helping patients make the initial lifestyle changes needed to reduce their risks, but patients often struggle to maintain those changes.

In this study the investigators propose to develop a novel mHealth application for supporting maintenance of physical activity. Kaiser Permanente Washington Health Research Institute (KPWHRI) will conduct a prospective study to test the application among Kaiser Permanente Washington (KPW) men and women with blood pressure that falls in the stage 1 hypertension range. By taking advantage of the frequent interactions that individuals have with their mobile phones throughout the day, the investigators will design and evaluate an adaptive, personalized application that (1) keeps patients reminded of their health goals and motivations; (2) provides actionable ideas for how patients can be active right now, given their current context; and (3) helps patients plan and reflect on their physical activity to enable creation of robust and sustainable physical-activity habits. In addition, the application will adapt its functioning for each patient over time in order to minimize user burden while optimizing its ability to encourage physical activity and maintain engagement with the intervention.

Through three Specific Aims-intervention development, intervention optimization, and pilot evaluation-this project will contribute: (1) understanding of how burden and intervention engagement change over time and how they are influenced by intervention delivery and patients' behavior and context; (2) generalization of learning algorithms that are used to personalize web content based on users' characteristics and past behavior for use in mHealth interventions for behavioral maintenance; and (3) new insights about how reflective and automated self-regulatory processes interact over time to support behavioral maintenance and how to optimally recruit these processes through an mHealth intervention.

Aim 2: Optimize intervention and investigate influences on participant response.

The investigators will conduct a three-month micro-randomized pilot study within-subject field study with 40-50 participants with blood pressure readings that fall in the stage 1 hypertension range. Goals for this aim include (1) perform in-situ usability and user-experience testing of the intervention; (2) finalize and tune the intervention's learning algorithms; (3) develop initial decision rules for when and for whom individual intervention components will be provided; and (4) begin to investigate how participants' physical activity, burden, and patterns of engagement with the intervention are affected by different intervention features and the context of use.

Aim 3: Pilot the personalized just-in-time adaptive mHealth intervention over 9 months The investigators will conduct a 9 month-long single-arm pilot study of adaptive mHealth intervention for physical-activity maintenance with 50-60 participants with blood pressure readings that falls in the stage 1 hypertension range. The investigators will (1) evaluate the feasibility and acceptability of the intervention for use over the course of nine months; (2) assess the ability of the learning algorithms to personalize intervention delivery over time; and (3) investigate how cardiac patients' responses to the intervention-physical activity, burden, and engagement-change over time as functions of time-varying application use and time-varying contextual factors. The study will also enable the investigators to gather empirical evidence to plan a follow-up RCT to test the efficacy of the intervention. Development of effective mHealth interventions requires advancements in and collaboration between computer science, human-computer interaction, and behavioral and health sciences. This project makes contributions to all three disciplines and deepens understanding of how to design personalized, adaptive interventions that help individuals not only to adopt but also sustain health-promoting behavior changes over the long-term.

Aim 2 and Aim 3 activities will take place sequentially. The recruitment and participant experience will be almost identical. Differences beyond scientific objectives between the Aim 2 and Aim 3 groups is the time each group is enrolled in the testing trial. Slight modifications are made to materials due to the difference in enrollment time.

No hypotheses will be tested. The purpose of both studies is to develop and test for usability and acceptability of an mHealth application that supports maintenance of physical activity of patients with high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Recent blood pressure readings that falls in the stage 1 hypertension range by new AHA/ACC guidelines [>= 130 systolic]
* Owns an iPhone
* Able to walk for 10 minutes without pain
* Expresses desire during study screen to increase physical activity

Exclusion Criteria:

* Taking hypertension meds
* Any diagnosis where physical activity would be counterindicated
* Recent acute cardio vascular event
* Major psychiatric illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
30 minute step count | 30 minutes
  step count within the 30-minute window after each available decision point when activity suggestions are randomized. Assessed using the Fitbit Versa Activity tracker.
Daily step count | 24 hours
  Daily step count on the day of treatment. Assessed using the Fitbit Versa activity tracker.

SECONDARY OUTCOMES:
MVPA | 24 hours
  Number of minutes of moderate or vigorous physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Pedja V Klasnja, PhD, Principal Investigator — Kaiser Permente Washington Health Research Institute
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset (i.e., containing no raw location/GPS information) will be generated and made available to the research community. The dataset will be stripped of all codes or any other information that could be linked back to the original data or to an individual participant. Prospective users of this dataset must agree to a confidentiality agreement, meaning that they must get permission from the HeartSteps Primary Investigator to share the data with anyone else. All external requests for data will be directed to Dr. Predrag Klasnja. Prospective investigators will submit a written proposal to the HeartSteps Investigator Team outlining the question they will investigate, the specific variables that they need to answer that question, their analytic plan for answering that question, and documentation of sufficient Institutional Review Board oversight (e.g., approval or exemption). Investigators will also need to sign a confidentiality agreement.
Supporting Information: Study Protocol